CLINICAL TRIAL: NCT06930456
Title: Intravenous Hydrocortisone Versus Ondansetron in Prevention of Post Spinal Anesthesia Hypotension in Elective Surgeries
Brief Title: Comparison Between Intravenous Hydrocortisone and Ondansetron in Prevention of Post Spinal Anesthesia Hypotension
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nada kamel Elgamal (Other)
Responsible Party: Sponsor-Investigator, Nada kamel Elgamal, Assistant Lecturer of Anesthesia and ICU, Port Said University hospital
Organization: Port Said University hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MED(3/12/2023)/(121)ANE921_002
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Post Spinal Anaesthesia Hypotension
MeSH Terms: interventions — Hydrocortisone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydrocortisone (H) group (Active Comparator): As in intervention description
  Interventions: Drug: hydrocortisone
- Ondansetron (O) group (Active Comparator): As in intervention description
  Interventions: Drug: ondansetron
- control (C) group (Placebo Comparator): As in intervention description
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hydrocortisone — A deidentified syringe (10 mL) containing 100 mg hydrocortisone will be given 15 minutes prior subarachnoid blockade. Spinal anesthesia will be performed with a 25-gauge Quincke spinal needle to administer 3.5 ml of a 0.5% hyperbaric bupivacaine plus 25 micrograms of fentanyl at the L3-L4 or L4-L5 level. Then, Patient will lie supine with slight head elevation. Intravenous Infusion of 500 ml normal saline over the initial post spinal 30 minutes. Sensory level and motor block will be verified. Heart rate (HR), systolic (SBP), diastolic (DBP) and mean blood pressure (MBP) will be measured every 5 min for 6 readings during which the patient remains in the supine position with no application of torniquet.
  Arms: Hydrocortisone (H) group
Drug: ondansetron — A deidentified syringe (10 mL) containing 8 mg ondansetron will be given 15 minutes prior subarachnoid blockade. Spinal anesthesia will be performed with a 25-gauge Quincke spinal needle to administer 3.5 ml of a 0.5% hyperbaric bupivacaine plus 25 micrograms of fentanyl at the L3-L4 or L4-L5 level. Then, Patient will lie supine with slight head elevation. Intravenous Infusion of 500 ml normal saline over the initial post spinal 30 minutes. Sensory level and motor block will be verified. Heart rate (HR), systolic (SBP), diastolic (DBP) and mean blood pressure (MBP) will be measured every 5 min for 6 readings during which the patient remains in the supine position with no application of torniquet.
  Arms: Ondansetron (O) group
Drug: Placebo — A deidentified syringe (10 mL) containing sterile distilled water for intravenous injection will be given 15 minutes prior subarachnoid blockade. Spinal anesthesia will be performed with a 25-gauge Quincke spinal needle to administer 3.5 ml of a 0.5% hyperbaric bupivacaine plus 25 micrograms of fentanyl at the L3-L4 or L4-L5 level. Then, Patient will lie supine with slight head elevation. Intravenous Infusion of 500 ml normal saline over the initial post spinal 30 minutes. Sensory level and motor block will be verified. Heart rate (HR), systolic (SBP), diastolic (DBP) and mean blood pressure (MBP) will be measured every 5 min for 6 readings during which the patient remains in the supine position with no application of torniquet.
  Arms: control (C) group

SUMMARY:
The purpose of this study is to assess and contrast the effectiveness of intravenous ondansetron and intravenous hydrocortisone in avoiding spinal anesthesia-induced hypotension.

DETAILED DESCRIPTION:
According to the medication investigated in this study, patients will be divided into three equal groups (40 each). Patients will receive one of the following 15 minutes before spinal anesthesia:

1. Hydrocortisone 100 mg (H group)
2. Ondansetron 8 mg (O group)
3. An identical volume of sterile distilled water (Control group) (C group).

Spinal anesthesia will be performed under complete aseptic conditions with the patient seated, a 25-gauge Quincke spinal needle is used to administer 3.5 ml of a 0.5% hyperbaric bupivacaine together with 25 micrograms of fentanyl at the L3-L4 or L4-L5 level.

Patients will lie supine with slight head elevation after the intrathecal injection is finished. Intravenous Infusion of 500 ml normal saline over the initial post spinal 30 minutes. Sensory level and motor block will be verified. Heart rate (HR), systolic (SBP), diastolic (DBP) and mean blood pressure (MBP) will be measured every 5 min for 30 min during which the patient remains in the supine position with no application of torniquet.

If the MAP drops by 20% below baseline or the systolic blood pressure falls below 90 mmHg, hypotension is recorded and will be treated with intravenous incremental doses of 5 mg ephedrine.

If the heart rate drops below 50 beats per minute, bradycardia is recorded, and atropine 0.5 mg will be administered intravenously. If ephedrine or atropine were used, only data from before their administration would be analyzed. The doses of ephedrine and atropine needed will be recorded.

Nausea, vomiting and shivering will be recorded when occur till the end of operation.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I and II (physical status according to American Society of Anesthesiologists).
2. Patients aged 21 years or more.
3. Either sex.
4. Abdominal and lower limb operations.

Exclusion Criteria:

1. Patient refusal.
2. hemodynamic instability
3. Hematological diseases, bleeding or coagulation abnormality.
4. Local skin infection and sepsis at site of spinal anesthesia
5. neuromuscular diseases (as myopathies, myasthenia gravies…)
6. Preexisting neurological deficit or psychiatric diseases.
7. Known intolerance to the study drugs.
8. patients already receiving any of the study drugs.
9. diabetic patient.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
hypotension | 5 minutes after subarachnoid injection and every 5 minutes for 30 minutes-duration
  The percentage of patients experiencing hypotension (a 20% decrease of the basal mean arterial blood pressure or systolic blood pressure less than 90 mmHg) at any point in the first thirty-minute period following spinal anesthetic induction

SECONDARY OUTCOMES:
bradycardia | 5 minutes after subarachnoid injection and every 5 minutes for 30 minutes-duration
  The percentage of patients experiencing bradycardia (HR less than 50 beat/min) at any point in the first thirty-minute period following spinal anesthesia.
requirement of atropine or ephedrine | 5 minutes after subarachnoid injection and every 5 minutes for 30 minutes-duration
  The proportion of those who require atropine or ephedrine for management of bradycardia or hypotension
Doses of administered atropine and ephedrine | 5 minutes after subarachnoid injection and every 5 minutes for 30 minutes-duration
  Doses of administered atropine and ephedrine
nausea and vomiting | after subarachnoid injection till the end of operation
  Incidence of post spinal nausea and vomiting till the end of operation
shivering | after subarachnoid injection till the end of operation
  Incidence of post spinal shivering till the end of operation
blood pressure and heart rate variations | 5 minutes after subarachnoid injection and every 5 minutes for 30 minutes-duration
  Variations in blood pressure and Heart Rate (HR).

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Ali Omera, prof. of Anesthesia and ICU, Study Chair — Port Said University, Faculty of Medicine, Department of Anesthesia
Locations (1):
- Port Said Hospital, Port Said, Port Said Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided